CLINICAL TRIAL: NCT01991379
Title: A Phase Ib/II Study of MEK162 in Combination With Imatinib Mesylate in Patients With Untreated Advanced Gastrointestinal Stromal Tumor (GIST)
Brief Title: MEK162 in Combination With Imatinib Mesylate in Patients With Untreated Advanced Gastrointestinal Stromal Tumor (GIST)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-162
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Stromal Tumor (GIST)
Keywords: MEK162; Imatinib; 13-162
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — binimetinib; Imatinib Mesylate; Blood Specimen Collection; Biopsy

ARMS (1):
- MEK162 in Combination With Imatinib Mesylate (Experimental): Pts will be treated with the combination therapy of MEK162 & imatinib. The phase Ib portion of the study, pts will receive imatinib at 400 mg once daily & MEK162 at the standard 3+3 escalation doses. Phase Ib expansion cohort, pts will receive the RP2D: imatinib 400 mg once daily (standard of care first line imatinib dose) & MEK162 at the RP2D twice daily. The phase II portion of the study, pts will receive imatinib at 400 mg once daily & MEK162 at the RP2D. The MEK162 RP2D was originally determined based on the phase Ib escalation data & it was established as 45 mg BID. After the completion of the phase Ib dose expansion & initiation of phase II, the MEK162 RP2D was reduced to 30 mg BID30 for better long term tolerability. Patient's will now begin MEK162 at the revised RP2D of 30 mg BID. 1 cycle is 28 days. If no progression of the tumor is seen, pts will continue on therapy. Pts who have progression of disease will proceed directly to second line therapy as per standard of care.
  Interventions: Drug: MEK162; Drug: Imatinib Mesylate (Gleevec®; STI571; NSC #716051); Other: Blood draws; Procedure: biopsy

INTERVENTIONS:
Drug: MEK162 — Patients should take the study drug with a glass of water. MEK162 can be taken with or without food.
Drug: Imatinib Mesylate (Gleevec®; STI571; NSC #716051)
Other: Blood draws
Procedure: biopsy — Following informed consent, the first 20 mandatory patients, except for patients who have already been treated with imatinib prior to consent, and subsequent voluntary patients enrolled on the phase II portion of the trial will undergo research biopsies. Patients should hold both imatinib and MEK162 doses on the day they undergo a biopsy.

SUMMARY:
The purpose of this study is to evaluate the effects, good and/or bad, of MEK162 and imatinib on the patient and on Gastrointestinal Stromal Tumor (GIST).

Funding Source - FDA OOPD, Array/Pfizer

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed GIST.
* In the Phase Ib portion, must have locally advanced or metastatic GIST and have progressed on imatinib.
* In the Phase II portion, patients must be newly diagnosed or treatment naïve, or have been off adjuvant imatinib therapy for at least 3 months. Patients with newly diagnosed GIST and who had been on imatinib for up to 4 weeks prior to signing the consent are allowed to enroll in order to expedite accrual.
* Patients must be at least 18 years of age.
* Disease must be measurable by RECIST 1.1.
* ECOG Performance Status 0 or 1.
* Adequate renal, hepatic, and hematologic function as the following: Serum Creatinine ≤ 1.5 mg/dL, Total Serum Bilirubin ≤ 1.5 x upper limit of normal (ULN), Serum AST (SGOT) and/or ALT (SGPT) ≤ 2.5 x ULN (or ≤ 5.0 x ULN if considered due to tumor)ANC ≥ 1500/mm3, Platelets ≥ 100,000/mm3, and hemoglobin ≥ 10g/dL.
* Patients of childbearing potential must have a negative serum pregnancy test within 14 days of treatment. Patients must agree to use a reliable barrier method of birth control during and for 3 months following the last dose of study drug.
* Patient must have adequate cardiac function (left ventricular ejection fraction (LVEF) ≥50% as determined by a multigated acquisition (MUGA) scan or echocardiogram; and QTc interval≤480 ms.
* Patient must be able to take oral medications.
* Patients must sign an informed consent document.

Exclusion Criteria:

* In the phase II portion of the study, patients that have been previously treated with any systemic therapy for GIST are not permitted to enroll, with the exception of adjuvant imatinib systemic therapy or exposure to imatinib within 4 weeks of signing consent.
* Patients have a severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
* Patients have known brain metastasis.
* Patients have known chronic liver disease (i.e., cirrhosis)
* Known positive serology for HIV, active Hepatitis B, and/or active Hepatitis C infection.
* Other active malignancy (other than malignancies, which the investigator determines are unlikely to interfere with treatment and safety analysis).
* Patients have a history or current evidence of Central Serous Retinopathy (CSR) or retinal vein occlusion (RVO) or predisposing factors to CSR or RVO (i.e. uncontrolled glaucoma or ocular hypertension, uncontrolled diabetes mellitus, hyperviscosity or hypercoagulability syndromes).
* History of retinal degenerative disease.
* History of Gilbert's syndrome.
* Patients have clinically significant cardiovascular disease, including any of the following:

  1) History of acute coronary syndrome including myocardial infarction, unstable angina, CABG, coronary angioplasty or stenting < 6 months prior to screening; 2) symptomatic chronic heart failure (New York Heart Association Criteria, Class II-IV); 3) evidence of clinically significant cardiac arrhythmias and/or conduction abnormalities < 6 months prior to screening except atrial fibrillation (AF) and paroxysmal supraventricular tachycardia (PSVT).
* Uncontrolled arterial hypertension despite appropriate medical therapy.
* Patients who have neuromuscular disorders that are associated with elevated creatinine phosphokinase (i.e. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
* Uncontrolled impairment of gastrointestinal function or gastrointestinal disease (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome). Patients who have ulcerative colitis or other gastrointestinal diseases that are well controlled are allowed to proceed with this study.
* Prior therapy with a MEK inhibitor.
* Patients had a major surgery within 3 weeks prior to study entry or who have not recovered from side effects of such procedure.
* Women who are pregnant or lactating.
* Sexually active males unless they use a condom during intercourse while taking the drug and for 15 days after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
* Patients with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-11; Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) (phase 1b portion) | 1 year
  The first three patients will be enrolled at Dose Level 1. If dose level 1 is not found to be tolerable, then the next cohort will be enrolled at dose level -1. If dose level -1 is not found to be tolerable, then the study may be terminated based on discussions with the sponsor and the combination may be deemed intolerable. If 0/3 patients or 1/6 patients experience a DLT on dose level 2, this will be the RP2D.
Best Response Rate (phase II portion) | 2 years
  Response Rate (CR+PR, RECIST 1.1). Response rate (RECIST 1.1) will be determined as the proportion of evaluable patients who have complete response or partial response defined by the RECIST 1.1.

SECONDARY OUTCOMES:
Response Rate (RR) (phase 1b portion) | 1 year
  defined by RECIST 1.1 criteria and by CHOI criteria RR will be estimated as the proportion of patients who have complete response or partial response for each criterion.
Progression Free Survival (PFS) | 1 year
  PFS will be calculated using Kaplan-Meier estimate among all patients enrolled. Patients who have not experienced the event of interest by the end of the study will be censored at the time of the last follow-up.
RR by CHOI criteria (phase II portion) | 1 year
  It will be determined as the proportion of patients who have complete response or partial response defined by the CHOI criteria with a two-sided 95% CI provided.
RR by EORTC criteria | 1 year
  It will be determined as the proportion of patients who have complete response or partial response defined by the EORTC criteria with a two-sided 95% CI provided.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Chi, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Chi P, Qin LX, Nguyen B, Kelly CM, D'Angelo SP, Dickson MA, Gounder MM, Keohan ML, Movva S, Nacev BA, Rosenbaum E, Thornton KA, Crago AM, Yoon S, Ulaner G, Yeh R, Martindale M, Phelan HT, Biniakewitz MD, Warda S, Lee CJ, Berger MF, Schultz ND, Singer S, Hwang S, Chen Y, Antonescu CR, Tap WD. Phase II Trial of Imatinib Plus Binimetinib in Patients With Treatment-Naive Advanced Gastrointestinal Stromal Tumor. J Clin Oncol. 2022 Mar 20;40(9):997-1008. doi: 10.1200/JCO.21.02029. Epub 2022 Jan 18. PMID 35041493
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/